CLINICAL TRIAL: NCT01078480
Title: Conservative Treatment Versus Plate Osteosynthesis Using Angular Stabile Screws and Precontoured Plates in Displaced Midshaft Clavicular Fractures. A Prospective Randomized Multicenter Study
Brief Title: Conservative Treatment Compared to Osteosynthesis in Patients With a Fractured Collar Bone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Collaborators: Central Jutland Regional Hospital (Other); Vejle Hospital (Other); Randers Regional Hospital (Other); Swemac Orthopaedics ApS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ON-001-CMJ
Record Dates: First submitted 2010-02-27; First posted 2010-03-02 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Displaced Midshaft Fracture of the Collar Bone
Keywords: Fracture; Collar bone
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm sling treatment (Experimental): Displaced midshaft fracture of the collar bone treated with an arm sling
  Interventions: Procedure: Displaced midshaft fracture of the collar bone
- Operation (Experimental): Displaced midshaft fracture of the collar bone treated with operation using a pre contoured titanium plate and screws.
  Interventions: Procedure: Operation using a precontoured titanium plate and screws

INTERVENTIONS:
Procedure: Operation using a precontoured titanium plate and screws — Operation using a precontoured titanium plate and screws
  Other Names: No other names.
  Arms: Operation
Procedure: Displaced midshaft fracture of the collar bone — Displaced midshaft fracture of the collar bone treated with an arm sling
  Other Names: No other names.
  Arms: Arm sling treatment

SUMMARY:
This study will compare non-operative treatment of displaced midshaft collarbone fractures with operative treatment using a precontoured titanium plate and screws.

The study hypothesis is that operation will provide better pain relief, faster return to activities, better function of the involved upper limb, and lower the risk of a non healing fracture (non union).

ELIGIBILITY:
Inclusion Criteria:

* fracture located to the mid third of the collar bone where there is no contact between the fractured surface of the main fragments on x-ray in one or two of two levels.

Exclusion Criteria:

* bilateral fracture
* imminent skin perforation
* open fracture
* associated neurovascular effect
* unstable fracture of neck of scapula "floating shoulder"
* fracture of coincidental upper extremity distal for the shoulder
* pathologic fracture
* the patient states that there was a unilateral or bilateral shoulder problem before the fracture
* fracture realized more than 14 days after it arose
* circumstances which make it impossible to carry out one of the two regimes, i.e. mental illness and abuse
* circumstances which make follow-up impossible, i.e. address far from the including departments and stays abroad of long duration
* medical contraindication against surgery or general anaesthesia
* former participation in the trial
* former fracture contra/ipsilateral at the age of 15 or older

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2010-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand (DASH) Score | 6 weeks, 3 months, 6 months, 1 year
  The DASH Outcome Measure is a 30-item, self-report questionnaire designed to measure physical function and symptoms in people with any of several musculoskeletal disorders of the upper limb. The tool gives clinicians and researchers the advantage of having a single, reliable instrument that can be used to assess any or all joints in the upper extremity.

SECONDARY OUTCOMES:
Constant-Murley Score | 6 weeks, 3 months, 6 months, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Carsten M Jensen, M.D.Sci., Principal Investigator — Orthopaedic Division, Central Jutland, Randers Hospital, Denmark
Locations (1):
- Orthopaedic Division, Randers Hospital, Randers, Central Jutland, Denmark

REFERENCES:
- [Derived] Qvist AH, Vaesel MT, Jensen CM, Jakobsen T, Jensen SL. Minimal Pain Decrease Between 2 and 4 Weeks After Nonoperative Management of a Displaced Midshaft Clavicle Fracture Is Associated with a High Risk of Symptomatic Nonunion. Clin Orthop Relat Res. 2021 Jan 1;479(1):129-138. doi: 10.1097/CORR.0000000000001411. PMID 32675585